CLINICAL TRIAL: NCT02048878
Title: Multi-Level Assessment of Physiologic Hyper-Arousal in Chronic Primary Insomnia: A Case Control Study
Brief Title: Hyper-Arousal in Chronic Primary Insomnia
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13-1214
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Chronic Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Insomnia group: Assessment of physiologic hyper-arousal across the two following domains:
  1. Sympathetic neural activity: recording at the level of the muscle by microneurography and at the level of the heart by spectral analysis of heart rate variability from the ECG signal obtained during sleep and wakefulness.
  2. Neurophysiologic arousal: recording of multiple sleep latency test (MSLT), recording of wake electroencephalography (EEG), and quantitative sleep EEG recording and analysis.
- Matched Control Group: Assessment of physiologic hyper-arousal across the two following domains:
  1. Sympathetic neural activity: recording at the level of the muscle by microneurography and at the level of the heart by spectral analysis of heart rate variability from the ECG signal obtained during sleep and wakefulness.
  2. Neurophysiologic arousal: recording of multiple sleep latency test (MSLT), recording of wake electroencephalography (EEG), and quantitative sleep EEG recording and analysis.

SUMMARY:
The purpose of this study is to determine whether individuals with chronic insomnia disorder have a higher degree of physiologic arousal (resulting in their trouble sleeping) than good sleepers. The primary goal is to perform a rigorous quantitative assessment of physiologic hyper-arousal across two domains (autonomic nervous system and neurophysiology) in patients with chronic primary insomnia as compared to good sleepers matched for sex, age, body mass index (BMI) and race/ethnicity.

ELIGIBILITY:
Inclusion Criteria for Insomniacs:

* Men and women with primary insomnia of at least 3 months in duration
* ages 21-65 years old
* BMI <35 kg/m2 to enable microneurography
* Moderate to severe insomnia based on the Insomnia Severity Index (ISI) questionnaire
* Pittsburgh Sleep Quality Index (PSQI) > 5
* Self-reported habitual sleep duration < 6.5 hours

Inclusion criteria for good sleepers:

* 21-65 years old men and women with BMI <35 kg/m2
* No insomnia based on ISI questionnaire
* Self-reported habitual sleep duration ≥ 6.5 hours but < 9 hours
* PSQI<5
* Sleep efficiency on PSG with TRT of 8 hours > 85%
* No history of mental illness, shift work, circadian rhythm disorders

Exclusion criteria for both insomniacs and good sleepers:

* Sleep disorders other than insomnia as assessed by screening PSG (apnea-hypopnea index or AHI ≥ 10, PLM arousal index ≥ 5)
* Circadian rhythm sleep disorders
* Diabetic based on HbA1c ≥ 6.5 %. For those with HbA1c ≥ 6.0 but <6.5%, the non-diabetic condition will be confirmed by 2-h oral glucose tolerance test
* History of meeting DSM-IVR criteria based on the Mini International Neuropsychiatric Interview version 6.0 for any major psychiatric disorder
* Unstable or serious medical conditions
* Current, or use within the past month, of psychoactive (other than stable treatment with antidepressants), hypnotic, stimulant or analgesic medications (except occasional non-narcotic analgesics), beta blockers or alpha blockers
* Shift work or other types of self imposed irregular sleep schedules
* Habitual smoking
* Habitual alcohol consumption
* Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Insomniacs and good sleepers
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, PhD, Principal Investigator — University of Chicago; Babak Mokhlesi, MD, Principal Investigator — University of Chicago; Jason R Carter, PhD, Principal Investigator — Michigan Technological University
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carter JR, Grimaldi D, Fonkoue IT, Medalie L, Mokhlesi B, Cauter EV. Assessment of sympathetic neural activity in chronic insomnia: evidence for elevated cardiovascular risk. Sleep. 2018 Jun 1;41(6):zsy048. doi: 10.1093/sleep/zsy048. PMID 29522186

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insomnia Group | Matched Control Group
Started | 13 | 15
Completed | 12 | 12
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insomnia Group | Matched Control Group | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (15) | 35 (13) | 37.3 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Sympathetic Baroreflex Sensitivity (BRS) Unit
Description: Direct recording of sympathetic nervous activity in a nerve of the lower leg using a micro-electrode.
Time Frame: 2 months after enrollment
Measure: Mean (Standard Deviation); unit: bursts per 100 heart beats per mm Hg
Arm/Group | Insomnia Group | Matched Control Group
Number analyzed (Participants) | 12 | 12
bursts per 100 heart beats per mm Hg | -2.1 (1.0) | -4.3 (1.3)

2. Primary Outcome: Systolic Arterial Pressure Reactivity
Description: Increase in blood pressure to stress
Time Frame: within 2 months after enrollment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Insomnia Group | Matched Control Group
Number analyzed (Participants) | 12 | 12
mmHg | 21 (11) | 14 (8)

3. Secondary Outcome: Multiple Sleep Latency Test (MSLT)
Description: MSLT will be used to objectively quantify tendency to fall asleep (sleep latency).
Time Frame: 2 months of enrollment
Population: One insomnia subject and one good sleeper control could not remain in the laboratory for the entire duration of the test due to personal scheduling issues.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Insomnia Group | Matched Control Group
Number analyzed (Participants) | 11 | 11
minutes
  Nap 1 | 8.7 (6.8) | 11.2 (8.2)
  Nap 2 | 7.3 (7.2) | 9.4 (6.1)
  Nap 3 | 6.8 (6.9) | 5.3 (3.2)
  Nap 4 | 6.7 (5.7) | 6.5 (6.4)
  Nap 5 | 12.7 (7.1) | 8.4 (7.1)

4. Secondary Outcome: Heart Rate Variability During Wake and During Sleep
Description: The balance between sympathetic and parasympathetic nervous control of the heart will be determined by spectral analysis of heart rate variability using continuous electrocardiogram (ECG) recording for 24 hours, including the normal sleep period.
Time Frame: 2 months after enrollment
Population: The biological signals were recorded but not submitted to the labor-intensive spectral analysis due to end of funding. Summary data were not generated. Therefore, no results on this outcome can be reported.
Arm/Group | Insomnia Group | Matched Control Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Electroencephalography (EEG) During Wake and Sleep
Description: The EEG will be measured continuously during sleep and at frequent intervals during wake. The signal will be submitted to power spectral analysis to examine spectral power in frequency bands that are typical of arousal and in frequency bands that are typical of deep sleep.
Time Frame: 2 months of enrollment
Population: as for outcome 4
Arm/Group | Insomnia Group | Matched Control Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Noninvasive Beat-to-beat Blood Pressure Monitoring
Time Frame: 2 months after enrollment
Population: Two insomnia subjects and 3 control subjects dropped out of the study after completing their first inpatient visit due to scheduling conflicts related to their professional occupation.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Insomnia Group | Matched Control Group
Number analyzed (Participants) | 10 | 9
mm Hg
  Systolic Blood Pressure dipping | 7.3 (11.9) | 15.2 (7.3)
  Diastolic Blood Pressure dipping | 3.0 (5.9) | 6.4 (2.5)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Insomnia Group | Matched Control Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No